CLINICAL TRIAL: NCT06415747
Title: Early Pain Finding in Infants With Brachial Plexus Birth Injury
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Kıvanç Delioğlu, Assistant Professor, Hacettepe University
Other Study IDs: GO 23/12
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Brachial Plexus Palsy
MeSH Terms: interventions — X-Rays

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Brachial Plexus Birth Injury: It was determined that 76 babies with BPBI and their families applied to our hospital for their first medical check or examination. Inclusion criteria: a diagnosis of BPBI, initial evaluation and not having started treatment before, being in the age range of 15-90 days old, and consent to participate in the study. Exclusion criteria: Children with BPBI who are older than 90 days or younger than 15 days and have started regular physical therapy or home program before applying to our hospital. In addition, causes of pseudo-paralysis that are diseases that may show symptoms similar to BPBI were excluded. Seventeen children who were excluded because they did not meet the inclusion criteria. Hence, 59 children with BPBI were included in the study.
  Interventions: Other: Observational pain and motor function assessments, and also comorbidities assessments with x-ray.

INTERVENTIONS:
Other: Observational pain and motor function assessments, and also comorbidities assessments with x-ray. — There was no intervention in our study, only observational and quantitative clinical evaluations.

SUMMARY:
In Brachail Plexus Birth Palsy (BPBI), fractures, glenohumeral joint dislocation, torticollis and plagiocephaly, facial nerve palsy, phrenic nerve palsy, obesity, speech delay, integumentary system problems, and central nervous system disorders are common comorbidities. Clinical assessments such as observation, palpation, and radiologic imaging are commonly used to identify early period comorbidities after delivery .Since fractures or joint deformities may occur in the affected upper extremity due to high-energy trauma at birth, pain assessment in the early postnatal period is recommended and several objective assessment methods have been proposed. Due to the difficulty of pain assessment in early childhood, the assessment is mostly performed by palpation. Pain is suspected if the baby grimaces with light palpation of the neck and upper shoulder area.

Although some hospitals have adopted objective assessment of pain and objective assessment is recommended, the level of pain in early childhood has not been investigated. Therefore, the aim of our study was to determine the level of pain in BPBI in early childhood and to examine the relationship between pain and motor function. In addition, the second aim of the study is to determine the cut-off value of the pain level that may be a sign of fracture in patients with BPBI, in order to suspect a fracture in the shoulder region and request additional examinations.

The diagnosis of BPBI, determination of Narakas classification and evaluation of comorbidities were performed by a senior orthopedic surgeon. After the initial doctor's examination, patients are routinely referred to the physiotherapy clinic for a physiotherapy evaluation.In the assessment, active joint movement and pain assessments of children were used, and all of these assessments were performed by a hand and pediatric physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* Having diagnosis of Brachial Plexus Birth Injury (BPBI),
* Being initial evaluation and not having started treatment before,
* Being in the age range of 15-90 days old,
* Consent to participate in the study.

Exclusion Criteria:

* Children with BPBI who are older than 90 days or younger than 15 days,
* Starting regular physical therapy or home program before applying to our hospital,
* Pseudo-paralysis that are diseases that may show symptoms similar to BPBI (clavicle or humerus fracture only, pseudo-paralysis not BPBI injury, glenohumeral joint septic arthritis, arthrogryposis multiplex congenita (AMC), cerebral palsy, spinal cord ischemic injury, spinal cord congenital aplasia, spinal tumor, congenital radial palsy).

Ages: 15 Days to 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: -In retrospective data collection, it was determined that 76 babies with BPBI and their families applied to our hospital for their first medical check or examination. Inclusion criteria were as follows: a diagnosis of BPBI, initial evaluation and not having started treatment before, being in the age range of 15-90 days old, and consent to participate in the study. Exclusion criteria: Children with BPBI who are older than 90 days or younger than 15 days and have started regular physical therapy or home program before applying to our hospital. Seventeen children who were excluded because they did not meet the inclusion criteria (4 had started physiotherapy or a home program, 1 had humerus fracture without BPBI, 1 had congenital radial palsy, 2 had AMC, 1 had spinal tumor, 8 were older than 90 days). Hence, 59 children with BPBI were included in the study.
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Comorbidities | Baseline, initial examination of children with BPBI who applied for medical follow-up.
  In BPBI, fractures, glenohumeral joint dislocation, torticollis and plagiocephaly, facial nerve palsy, phrenic nerve palsy, obesity, speech delay, integumentary system problems, and central nervous system disorders are common comorbidities. In our university hospital, humerus or scapula fracture, glenohumeral joint dislocation, torticollis and plagiocephaly, facial nerve palsy, phrenic nerve palsy, Horner's syndrome, and central nervous system disorders are checked with clinical examinations and X-ray to record as a comorbidities and additional problems.
Active Movement Scale - Motor Function Assessment | Baseline, initial examination of children with BPBI who applied for medical follow-up.
  The AMS is a standardized assessment of 15 active joint movements on the affected side using an eight-point scale. The 15 movements were assessed by the AMS include. For each movement, the range of 0-4 points is evaluated in gravity eliminated position, while the range of 5-7 represents movement against gravity. The AMS-Total score is the sum of the scores of all 15 movements and represents the total function of the affected upper extremity, therefore the score can range from 0 to 105 points, with 0 being poor and 105 being the best score.
Flacc Pain Scale | Baseline, initial examination of children with BPBI who applied for medical follow-up.
  The FLACC Pain Scale is an observational behavioral scale developed by Merkel et al. in 1997. It provides a simple and consistent method for the assessment of pain in early childhood, especially in the age group when the child cannot verbally express his pain. It is used to evaluate procedural and postoperative pain in children older than 1 month. The FLACC scale is used to assess pain at rest, during a medical procedure or during various environmental stimuli. It scores 5 behaviors of the infant, including facial expression, leg movements, activities, crying and consolability, between 0 and 2 points. The scale produces a total pain score between 0 and 10 points.

CONTACTS AND LOCATIONS:
Overall Officials: Kıvanç Delioğlu, Assist Prof, Principal Investigator — Hacettepe University; Akin Uzumcugil, Assoc Prof, Study Chair — Hacettepe University; Ebru Ozturk, PhD, Study Chair — Hacettepe University; Mintaze Kerem, Professor, Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Faculty of Physical Therapy Rehabilitation, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No